CLINICAL TRIAL: NCT04273529
Title: The Efficacy and Safety of Thalidomide in the Adjuvant Treatment of Moderate New Coronavirus (COVID-19) Pneumonia: a Prospective, Multicenter, Randomized, Double-blind, Placebo, Parallel Controlled Clinical Study
Brief Title: The Efficacy and Safety of Thalidomide in the Adjuvant Treatment of Moderate New Coronavirus (COVID-19) Pneumonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Second Affiliated Hospital of Wenzhou Medical University (Other); Wenzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20200214-COVID-19-M-T
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: COVID-19 Thalidomide
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): placebo
  Interventions: Drug: placebo
- Thalidomide group (Experimental): thalidomide
  Interventions: Drug: thalidomide

INTERVENTIONS:
Drug: thalidomide — 100mg，po，qn，for 14 days.
  Other Names: fanyingting
  Arms: Thalidomide group
Drug: placebo — 100mg，po，qn，for 14 days.
  Arms: Control group

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (2019-nCoV) from these pneumonia patients and developed a real-time reverse transcription PCR (real time RT-PCR) diagnostic assay.

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Thalidomide has anti-inflammatory, anti-fibrotic, anti-angiogenesis, and immune regulation effects. This study is the first Prospective, Multicenter, Randomized, Double-blind, Placebo, Parallel Controlled Clinical Study at home and abroad to use immunomodulators to treat patients with COVID-19 infection.

DETAILED DESCRIPTION:
The new coronavirus (COVID-19) [1] belongs to the new beta coronavirus. Current research shows that it has 85% homology with bat SARS-like coronavirus (bat-SL-CoVZC45), but its genetic characteristics are similar to SARSr-CoV. There is a clear difference from MERSr-COV. Since December 2019, Wuhan City, Hubei Province has successively found multiple cases of patients with pneumonia infected by a new type of coronavirus. With the spread of the epidemic, as of 12:00 on February 12, 2020, a total of 44726 confirmed cases nationwide (Hubei Province) 33,366 cases, accounting for 74.6%), with 1,114 deaths (1068 cases in Hubei Province), and a mortality rate of 2.49% (3.20% in Hubei Province).

In view of the fact that there is currently no effective antiviral therapy, the prevention or treatment of lung injury caused by COVID-19 can be an alternative target for current treatment. Thalidomide has anti-inflammatory, anti-fibrotic, anti-angiogenesis, and immune regulation effects. In the early clinical practice of treating severe A H1N1, it was clinically concerned, and combined with hormones and conventional treatment, and achieved good results.

Although the death rate of COVID-19 infected persons is not high, their rapid infectiousness and the lack of effective antiviral treatment currently have become the focus of the national and international epidemic. Thalidomide has been available for more than sixty years, and has been widely used in clinical applications. It has been proved to be safe and effective in IPF, severe H1N1 influenza lung injury and paraquat poisoning lung injury, and the mechanism of anti-inflammatory and anti-fibrosis is relatively clear. As the current research on COVID-19 at home and abroad mainly focuses on the exploration of antiviral efficacy, this study intends to find another way to start with host treatment in the case that antiviral is difficult to overcome in the short term, in order to control or relieve lung inflammation caused by the virus To improve lung function. This study is the first study at home and abroad to use immunomodulators to treat patients with COVID-19 infection. It is hoped that the patients can get out of the bitter sea as soon as possible and provide effective solutions for the country and society.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Laboratory (RT-PCR) diagnosis of common patients infected with COVID-19 (refer to the fifth edition of the Chinese Guidelines for Diagnosis and Treatment);
3. chest imaging confirmed lung damage;
4. The diagnosis is less than or equal to 8 days;

Exclusion Criteria:

1. Severe liver disease (such as Child Pugh score ≥ C, AST> 5 times the upper limit); severe renal dysfunction (the glomerulus is 30ml / min / 1.73m2 or less)
2. Positive pregnancy or breastfeeding or pregnancy test;
3. In the 30 days before the screening assessment, have taken any experimental treatment drugs for COVID-19 (including off-label, informed consent use or trial-related);
4. Those with a history of thromboembolism, except for those caused by PICC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical recoveryTime to Clinical Recovery (TTCR) | up to 28 days
  TTCR is defined as the time (in hours) from initiation of study treatment (active or placebo) until normalisation of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 72 hours. Normalisation and alleviation criteria:
  Fever - ≤36.6°C or -axilla, ≤37.2 °C oral or ≤37.8°C rectal or tympanic, Respiratory rate - ≤24/minute on room air, Oxygen saturation - >94% on room air, Cough - mild or absent on a patient reported scale of severe, moderate, mild, absent.

SECONDARY OUTCOMES:
All cause mortality | up to 28 days
  baseline SpO2 during screening, PaO2/FiO2 <300mmHg or a respiratory rate ≥ 24 breaths per min without supplemental oxygen
Frequency of respiratory progression | up to 28 days
  Defined as SPO2≤ 94% on room air or PaO2/FiO2 <300mmHg and requirement for supplemental oxygen or more advanced ventilator support.
Time to defervescence | up to 28 days
  in those with fever at enrolment

OTHER OUTCOMES:
Time to cough reported as mild or absent | up to 28 days
  in those with cough at enrolment rated severe or moderate
Respiratory improvement time | up to 28 days
  patients with moderate / severe dyspnea when enrolled
Frequency of requirement for supplemental oxygen or non-invasive ventilation | up to 28 days
Time to 2019-nCoV RT-PCR negative in upper respiratory tract specimen | up to 28 days
Change (reduction) in 2019-nCoV viral load in upper respiratory tract specimen as assessed by area under viral load curve | up to 28 days
Frequency of requirement for mechanical ventilation | up to 28 days
Frequency of serious adverse events | up to 28 days
Serum TNF-α, IL-1β, IL-2, IL-6, IL-7, IL-10, GSCF, IP10，MCP1, MIP1α and other cytokine expression levels before and after treatment | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jinglin Xia, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University

REFERENCES:
- [Background] Zhao L, Xiao K, Wang H, Wang Z, Sun L, Zhang F, Zhang X, Tang F, He W. Thalidomide has a therapeutic effect on interstitial lung fibrosis: evidence from in vitro and in vivo studies. Clin Exp Immunol. 2009 Aug;157(2):310-5. doi: 10.1111/j.1365-2249.2009.03962.x. PMID 19604271
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Background] Jin YH, Cai L, Cheng ZS, Cheng H, Deng T, Fan YP, Fang C, Huang D, Huang LQ, Huang Q, Han Y, Hu B, Hu F, Li BH, Li YR, Liang K, Lin LK, Luo LS, Ma J, Ma LL, Peng ZY, Pan YB, Pan ZY, Ren XQ, Sun HM, Wang Y, Wang YY, Weng H, Wei CJ, Wu DF, Xia J, Xiong Y, Xu HB, Yao XM, Yuan YF, Ye TS, Zhang XC, Zhang YW, Zhang YG, Zhang HM, Zhao Y, Zhao MJ, Zi H, Zeng XT, Wang YY, Wang XH; , for the Zhongnan Hospital of Wuhan University Novel Coronavirus Management and Research Team, Evidence-Based Medicine Chapter of China International Exchange and Promotive Association for Medical and Health Care (CPAM). A rapid advice guideline for the diagnosis and treatment of 2019 novel coronavirus (2019-nCoV) infected pneumonia (standard version). Mil Med Res. 2020 Feb 6;7(1):4. doi: 10.1186/s40779-020-0233-6. PMID 32029004
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Wen H, Ma H, Cai Q, Lin S, Lei X, He B, Wu S, Wang Z, Gao Y, Liu W, Liu W, Tao Q, Long Z, Yan M, Li D, Kelley KW, Yang Y, Huang H, Liu Q. Recurrent ECSIT mutation encoding V140A triggers hyperinflammation and promotes hemophagocytic syndrome in extranodal NK/T cell lymphoma. Nat Med. 2018 Feb;24(2):154-164. doi: 10.1038/nm.4456. Epub 2018 Jan 1. PMID 29291352
- [Background] Kwon HY, Han YJ, Im JH, Baek JH, Lee JS. Two cases of immune reconstitution inflammatory syndrome in HIV patients treated with thalidomide. Int J STD AIDS. 2019 Oct;30(11):1131-1135. doi: 10.1177/0956462419847297. Epub 2019 Sep 19. No abstract available. PMID 31533530
- [Background] Zhu H, Shi X, Ju D, Huang H, Wei W, Dong X. Anti-inflammatory effect of thalidomide on H1N1 influenza virus-induced pulmonary injury in mice. Inflammation. 2014 Dec;37(6):2091-8. doi: 10.1007/s10753-014-9943-9. PMID 24912813
- [Result] Bartlett JB, Dredge K, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. Nat Rev Cancer. 2004 Apr;4(4):314-22. doi: 10.1038/nrc1323. No abstract available. PMID 15057291